CLINICAL TRIAL: NCT06956196
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Stapokibatrt in Children With Moderate-to-severe Atopic Dermatitis
Brief Title: Study of Stapokibatrt in Children Subjects With Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-101217
Record Dates: First submitted 2025-04-30; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stapokibatrt group (Experimental)
  Interventions: Biological: Stapokibatrt
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Stapokibatrt — Stapokibatrt 1 or 2 ml,Subcutaneous injection(SC)
  Arms: Stapokibatrt group
Other: Placebo — Placebo of matching volume，Subcutaneous injection(SC)
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled phase 3 study to evaluate the efficacy, safety, Pharmacokinetics(PK), PharmacoDynamics(PD) and immunogenicity of Stapokibatrt in children with moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 and ≤ 11 years old.
* Diagnosis of AD according to the American Academy of Dermatology Consensus (2014) Criteria.
* With moderate-to-severe AD, and inadequate response to topical medications.

Exclusion Criteria:

* Prior treatment with Stapokibart
* Treatment with dupilumab within 13 weeks prior to the baseline visit, or treatment with anti-IgE(Immunoglobulin E) monoclonal antibody，other biological agents within 5 half-lives prior to the baseline visit .
* Treatment with immunosuppressants/immunomodulatory drugs, ultraviolet therapy, or systemic traditional Chinese medicine for AD within 4 weeks prior to the baseline visit.
* Treatment with a topical corticosteroids (TCS), topical calcineurin inhibitor (TCI) or topical Phosphodiesterase-4(PDE-4) inhibitor within 1 weeks prior to the baseline visit.
* History of atopic keratoconjunctivitis invading cornea.
* Acute attacks of Atopic Dermatitis within 4 weeks prior to the baseline visit.
* Planned major surgical procedure during the patient's participation in this study.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving Eczema Area and Severity Index(EASI-75) at week 18 | Up to week 18
  The EASI is a composite index with scores ranging from 0 to 72. Four Atopic Dermatitis(AD) disease characteristics (erythema, edema/papulation, excoriation, lichenification) will each be assessed for severity by the investigator on a scale of "0" (none) through "3" (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ma, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital Capital Medical University, Beijing, China